CLINICAL TRIAL: NCT06236581
Title: Glycemic Excursion Minimization (GEM) to Outshine Health Disparities: RCT
Brief Title: Glycemic Excursion Minimization (GEM) to Outshine Health Disparities
Acronym: GEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catherine Davis (Other)
Collaborators: University of Virginia (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor-Investigator, Catherine Davis, Professor, Augusta University
Organization: Augusta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1974851
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Type 2 Diabetes
Keywords: Black; Continuous glucose monitoring; physical activity; carbohydrate
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, intervention vs. waitlist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GEM Intervention (Experimental): A lifestyle coach will deliver the GEM intervention over 4 weeks in person and/or virtually (synchronously) to permit interaction with participants. A pocket-sized manual will be provided with 4 units corresponding to session topics, and diary pages to record glucose responses to food and physical activity (PA). Session 1: Introduce GEM, identify personal motivation, learn about foods that cause glucose to go high (high glycemic load (GL) foods) and those that do not (low GL foods), learn how physical activity affects glucose, and begin monitoring how these choices affect glucose. Session 2: Replacement, substitution, and portion control to reduce consumption of high GL foods. Session 3: Increasing PA and reducing sedentary behavior, esp. after a meal. Session 4: Ways to continue lifestyle changes over a lifetime, handle relapses, and thank loved ones for their support. Text message reminders may be sent to participants between sessions to prompt diary entries and for encouragement.
  Interventions: Behavioral: GEM Intervention
- Waitlist (No Intervention): Participants will be invited to receive the GEM intervention after they posttest, the next time it is offered.

INTERVENTIONS:
Behavioral: GEM Intervention — Lifestyle coaching
  Arms: GEM Intervention

SUMMARY:
The purpose of this study is to see if the GEM intervention is acceptable and helpful to Black adults with type 2 diabetes. The GEM intervention (coaching to reduce carbohydrate intake and increase physical activity after meals, with feedback from a continuous glucose monitor, CGM) might improve blood glucose levels, reduce diabetes distress, and increase empowerment and confidence in managing diabetes.

DETAILED DESCRIPTION:
The purpose of the study is to test the feasibility, acceptability, and initial efficacy of the tailored GEM intervention among adult Black patients with type 2 diabetes, who are not on insulin or secretagogues.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* capable of making dietary and physical activity changes

Exclusion Criteria:

* on insulin or secretagogue
* on medications that impede weight loss (e.g., prednisone)
* pregnant or planning pregnancy in the next 2 months
* no history of moderate to severe hypoglycemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on percent time in range from continuous glucose monitor at post-intervention | Baseline week and post-intervention week. From baseline week to the week after end of intervention or waitlist period, up to 6 weeks
  Difference in percent of time in range (70-180 mg/dL) from continuous glucose monitor data. Change = post intervention week minus baseline week.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine L Davis, PhD, Principal Investigator — Augusta University
Locations (1):
- Georgia Prevention Institute, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
The small number of expected participants means there is too great a risk of loss of confidentiality. Group level data will be shared upon request to qualified researchers.